CLINICAL TRIAL: NCT03997188
Title: Study for the Evaluation of the Impact of HEPILOR on the Possible Delay in the Development of Dysphagia in Breast Cancer Patients Undergoing Adjuvant Radiotherapy on the Breast/Thoracic Wall and Lymph Node Drainage.
Brief Title: Zinc-L-Carnosine Prevents Dysphagia in Breast Cancer Patients Undergoing Adjuvant Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cynthia Aristei (Other)
Responsible Party: Sponsor-Investigator, Cynthia Aristei, Professor, University Of Perugia
Organization: University Of Perugia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003 (Hepilor)
Record Dates: First submitted 2019-06-05; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer Female; Dysphagia; Adjuvant Radiotherapy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: note Study Phase* A medical device is a substance; whose purpose is comparable to the drug ( therapy, prevention, diagnosis, restoration of functions), but it is different from the drug because the drug acts with pharmacological, metabolic and immunological means, while the medical device acts through a mechanical action. Hepilor is a medical device in the form of a syrup with specific properties to protect and repair the gastro-intestinal mucosa. The functional substances of the medical device (Zinc-L-Carnosine and Sodium Alginate) thanks to their mucoadhesive properties act as a physical barrier protecting the damaged areas. In consideration of this we have designed a randomized phase III to to determine whether ZLC prevented or delayed esophagitis in breast cancer patients undergoing HeT to SC/IC lymph nodes and residual breast or chest wall.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepilor arm (Experimental): patients received ZLC solution. The prescribed dose was 10 ml, in the morning and evening, between meals.
  Interventions: Device: Hepilor
- Placebo arm (Placebo Comparator): Patients received a placebo solution. The prescribed dose was 10 ml, in the morning and evening, between meals
  Interventions: Device: Hepilor

INTERVENTIONS:
Device: Hepilor — ZLC oral suspension and placebo were both started on Day 1 of RT-HeT and ended when RT was completed or at the onset of dysphagia.
  Other Names: Placebo

SUMMARY:
Irradiation of level III and IV draining nodes in breast cancer patients is often associated with dysphagia, requiring treatment with FANS and/or steroids. The present randomized phase III trial determined whether Zinc-L-Carnosine ( Hepilor), prevents or delays the onset of dysphagia in these patients.

DETAILED DESCRIPTION:
. This is a randomized phase III prospective placebo-controlled trial with patients recruited from one single university teaching hospital. Inclusion criteria were: age ≥18 years, breast cancer patients who were candidates for post-operative RT by means of HeT to the breast /chest wall and SC/IC nodes (III-IV levels).Exclusion criteria were: pregnancy or lactation, known or suspected hypersensitivity or allergy to ZLC or to any of the excipients in its oral solution.

All patients were randomized by a pre-determined computer code to two groups.

1. HEPILOR arm: patients received ZLC solution
2. Placebo arm: patients received a placebo solution Toxicity was assessed weekly in all patients immediately before or after the RT session. Acute toxicity was defined as occurring during RT or in 30 days after it ended and assessed using the Common Terminology Criteria for Adverse Events (CTCAE 4.0 scale). Dysphagia was assessed weekly by means of EAT 10, a self-administered questionnaire

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* breast cancer patients who were candidates for post-operative RT by means of HeT to the breast /chest wall and SC/IC nodes (III-IV levels).

Exclusion Criteria:

* pregnancy or lactation
* known or suspected hypersensitivity or allergy to ZLC or to any of the excipients in its oral solution.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Zinc-L-Carnosine prevents dysphagia in breast cancer patients undergoing adjuvant radiotherapy: clinical outcome assessed by Eating Assessment Tool (EAT-10) questionaire | once a week during the radiotherapy and once at first month of follow-up
  The Primary end-point was no dysphagia. The study aim is to assess whether the medical device is able to avoid or delay the onset of dysphagia. The patients were evaluated before the start of radiotherapy and weekly to identify the possible appearance of dysphagia. Dysphagia was assessed weekly by means of self-assessment EAT10 questionnaire that is a tool used to assess objectively the presence of dysphagia, in details (0 = No problem 4 = Severe problem): 1. My swallowing problem has caused me to lose weight; 2. My swallowing problem interferes with my ability to go out for meals; 3. Swallowing liquids takes extra effort; 4. Swallowing solids takes extra effort; 5. Swallowing pills takes extra effort; 6. Swallowing is painful; 7. The pleasure of eating is affected by my wallowing; 8. When I swallow food sticks in my throat; 9. I cough when I eat; 10. Swallowing is stressful.
Degree of dysphagia | only in the presence of dysphagia:once a week during the radiotherapy and once at first month of follow-up
  The degree of dysphagia was evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) 4.0 scale.
  When the patient showed a score of the questionnaire greater than 3 the target was reached dysphagia was present and this was evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Dysphagia =Grade 1: Symptomatic, able to eat regular diet. Grade 2: Symptomatic and altered eating/swallowing. Grade 3: Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aristei, MD, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No